CLINICAL TRIAL: NCT01051440
Title: A Magnetic Resonance Spectroscopy and fMRI Study of the Effects of Lisdexamfetamine on Bipolar Depression
Brief Title: Magnetic Resonance Imaging Study of Lisdexamfetamine for Bipolar Depression
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Slow enrollment
Sponsor: Steward St. Elizabeth's Medical Center of Boston, Inc. (Other)
Collaborators: Shire (Industry)
Responsible Party: Principal Investigator, Michael Henry, MD, Principal Investigator, Steward St. Elizabeth's Medical Center of Boston, Inc.
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 00517
Record Dates: First submitted 2010-01-14; First posted 2010-01-18 (Estimated); Results first posted 2013-01-30 (Estimated); Last update posted 2013-01-30 (Estimated); Status verified 2012-12

CONDITIONS: Bipolar Depression
Keywords: lisdexamfetamine; vyvanse; bipolar disorder; depression; stimulant; magnetic resonance spectroscopy; functional magnetic resonance imaging; neuropsychological testing
MeSH Terms: conditions — Bipolar Disorder; Depression | interventions — Lisdexamfetamine Dimesylate

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (2):
- Placebo (Placebo Comparator): Subjects will receive placebo for lisdexamfetamine.
  Interventions: Drug: Placebo
- Lisdexamfetamine (Active Comparator): Subjects will start with 20 mg per day of lisdexamfetamine and may increase to a maximum of 40 mg.
  Interventions: Drug: Lisdexamfetamine

INTERVENTIONS:
Drug: Lisdexamfetamine — Start at 20 mg daily. Increased to a maximum of 40 mg daily. Can be decreased in 10 mg increments.
  Other Names: Vyvanse
  Arms: Lisdexamfetamine
Drug: Placebo — Subjects will receive placebo matched to lisdexamfetamine.
  Arms: Placebo

SUMMARY:
There have been reports that stimulants may be effective for bipolar depression without triggering mania. This study will examine whether lisdexamfetamine can improve depressive symptoms over the course of eight weeks. Lisdexamfetamine is a prodrug stimulant that is currently approved for attention deficit hyperactivity disorder (ADHD). Participants take the study drug or placebo in addition to a mood stabilizer. The study includes functional magnetic resonance imaging and magnetic resonance spectroscopy to determine whether the medication alters the response to affective stimuli or glutamate, glutamine, or gamma aminobutyric acid (GABA) levels. Neuropsychological testing is also included to determine whether the study drug improves memory and attention in this population. The primary hypothesis is that lisdexamfetamine is clinically effective in this population. The secondary hypothesis is that it will result in an increased response to affective stimuli and altered neurotransmitter levels in the anterior cingulate cortex.

ELIGIBILITY:
Inclusion Criteria:

* Aged 21 to 50 years.
* Diagnosed with Bipolar Disorder I or II disorder.
* Currently in the depressive phase of the illness.
* Montgomery Asberg Depression Rating Scale (MADRS) score greater than 15.
* Medication regimen (Lamotrigine, Valproate, Lithium, either alone or in combination with atypical antipsychotics, or typical antipsychotics) at stable doses for at least one month.
* Has an established residence and phone.
* Capable of providing informed consent.

Exclusion Criteria:

* Met Diagnostic and Statistical Manual 4th edition (DSM-IV-TR) criteria for rapid cycling within the 6 months prior to enrolling in the study.
* Meets DSM-IV-TR criteria for Schizophrenia, Schizoaffective disorder, Post-Traumatic Stress disorder, Obsessive-Compulsive disorder, or Eating disorder. Co-morbid anxiety disorders are not a reason for exclusion.
* History of psychotic symptoms at any point during the subject's illness.
* Met DSM-IV-TR criteria for alcohol or substance (except for nicotine) dependence or abuse within the past 6 months.
* Lifetime history of amphetamine abuse or dependence.
* Subject has a lifetime history of stimulant-induced mania
* History of seizures, including febrile seizures in childhood.
* Young Mania Rating Scale (YMRS) greater than 8.
* History of significant coronary artery disease, angina, untreated or inadequately treated thyroid disease (less than 1 month chemically euthyroid), type I diabetes, autoimmune disease, glaucoma, hypertension, seizures, or other medical condition(s) which in the opinion of the principal investigator is likely to significantly impact the subject's mood or potential response to the study medication.
* Electrocardiogram (ECG) with significant arrhythmias or conduction abnormalities, which in the opinion of the physician investigator preclude study participation; uncontrolled hypertension (>160/100) or tachycardia (heart rate >110).
* Female subjects who are peri or post-menopausal.
* Subjects taking Ritalin or other stimulants, theophylline, steroids, atomoxetine, cholinesterase inhibitors, memantine, modafinil, warfarin, anticonvulsants, clonidine, theophylline, monoamine oxidase inhibitors, and pseudoephedrine, or other medications that are likely to significantly interact (either pharmacokinetically or pharmacodynamically) with the subject's mood or Lisdexamfetamine.
* Subject regularly (more than 4 days per week) ingests more than four caffeine containing drinks per day.
* Pregnancy.
* In women of childbearing potential, an unwillingness to avoid pregnancy for the duration of the study.
* Active suicidal ideation.
* History of homicidal ideation.
* Allergy or other clinical condition which prohibits the use of all of the approved mood stabilizers or Lisdexamfetamine.
* Metal in the body (e.g. history of working as a sheet metal worker) or pacemaker which is a contra-indication to magnetic resonance imaging (MRI).
* Significant claustrophobia.

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 2 (Actual)
Dates: Start 2010-02; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael E Henry, MD, Principal Investigator — Steward St. Elizabeth's Medical Center of Boston, Inc.
Locations (1):
- Steward St. Elizabeth's Medical Center, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The recruitment period began in June 2010 and concluded in early 2012. Recruitment was through media advertisements and patients in the hospital outpatient clinic. Out of hundreds of individuals who were pre-screened by telephone, 31 were invited to the clinic for screening visits.
Pre-assignment Details: Participants who were not on an approved mood stabilizer (lithium, valproate, or lamotrigine) at the time of enrollment were eligible for a one-month lead in to start a mood stabilizer prior to randomization. Several participants were excluded due to psychiatric co-morbidity, unclear diagnosis, history of stimulant use, or medical concerns.
Groups:
- Placebo: Subjects received matched placebo for lisdexamfetamine.
- Lisdexamfetamine: Subjects started with 20 mg per day of lisdexamfetamine and could have the dose increased to a maximum of 40 mg based on change in clinical response and adverse events.
Period: Overall Study
Arm/Group | Placebo | Lisdexamfetamine
Started | 1 | 1
Completed | 1 | 1
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Lisdexamfetamine | Total
Number analyzed (Participants) | 1 | 1 | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 1 | 2
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 38 (0) | 30 (0) | 34 (5.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Change in Montgomery Asberg Depression Rating Scale (MADRS) Score Over Time.
Description: The change in MADRS score from the baseline visit to the week 8 visit is reported. The MADRS is a clinician-rated scale that consists of 10 items rated on a from 0 to 6 (maximum score of 60), with higher scores indicating greater symptom severity. An increase in score indicates a worsening of symptoms whereas a decrease indicates an improvement in symptoms.
Time Frame: baseline and 8 weeks
Population: All participants randomized to lisdexamfetamine or placebo were included.
Measure: Number; unit: units on a scale
Arm/Group | Placebo | Lisdexamfetamine
Number analyzed (Participants) | 1 | 1
units on a scale | 4 (0) | -22 (0)

2. Secondary Outcome: Change in Clinical Global Impressions Severity (CGI-S) Score.
Description: The CGI-S score reflects the clinician's overall impression of the patient's functional status. The scoring for the single item ranges from 1 with an anchor of "normal, not at all ill" to 7 with an anchor of "among the most extremely ill patients". Thus, higher scores indicate greater severity of symptoms.
Time Frame: baseline and week 8
Population: All participants who were randomized to lisdexamfetamine or placebo were included.
Measure: Number; unit: units on a scale
Arm/Group | Placebo | Lisdexamfetamine
Number analyzed (Participants) | 1 | 1
units on a scale | 1 | -2

3. Secondary Outcome: Change in Clinical Global Impressions Improvement (CGI-I) Score.
Description: The CGI-I score indicates the clinician's overall assessment of improvement in function from one visit to the next. The single item is scored from 1 to 7 with anchor points ranging from very much improved (1) to very much worse (7). A decrease in score reflects an improvement in functional status.
Time Frame: week 1 and week 9
Population: All participants who were randomized to lisdexamfetamine or placebo were included.
Measure: Number; unit: units on a scale
Arm/Group | Placebo | Lisdexamfetamine
Number analyzed (Participants) | 1 | 1
units on a scale | 0 | -2

ADVERSE EVENTS:
Arm/Group | Placebo | Lisdexamfetamine
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/1
Other Adverse Events (participants affected / at risk) | 0/1 | 0/1

LIMITATIONS AND CAVEATS:
The study was terminated before completion due to low enrollment. One subject was randomized to lisdexamfetamine and one was randomized to placebo. Therefore, it was not possible to obtain complete data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No